CLINICAL TRIAL: NCT00690560
Title: International Phase II Study Evaluating the Association of CHOP-rituximab With Consolidation by Early Ibritumomab Tiuxetan-Y90 in Patients Aged 65 to 80 Years With CD20+ Large Cell Malignant Lymphoma and no Prior Therapy
Brief Title: Combination Chemotherapy, Rituximab, and Yttrium Y 90 Ibritumomab Tiuxetan in Treating Patients With Newly Diagnosed Large B-Cell Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Centre Antoine Lacassagne (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2006/27; CALACASS-3RCHOPZ; INCA-RECF0624; 2006-006179-19 (EudraCT Number); CALACASS-2006/27
Record Dates: First submitted 2008-06-03; First posted 2008-06-04 (Estimated); Last update posted 2025-09-30 (Actual); Status verified 2015-02

CONDITIONS: Lymphoma
Keywords: contiguous stage II adult diffuse large cell lymphoma; noncontiguous stage II adult diffuse large cell lymphoma; stage I adult diffuse large cell lymphoma; stage III adult diffuse large cell lymphoma; stage IV adult diffuse large cell lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, Large B-Cell, Diffuse | interventions — Rituximab; Cyclophosphamide; Doxorubicin; Prednisone; Vincristine; ibritumomab tiuxetan

ARMS (1):
- R-CHOP14 chemotherapy (Experimental)
  Interventions: Biological: rituximab; Drug: cyclophosphamide; Drug: doxorubicin hydrochloride; Drug: prednisone; Drug: vincristine sulfate; Radiation: yttrium Y 90 ibritumomab tiuxetan

INTERVENTIONS:
Biological: rituximab
Drug: cyclophosphamide
Drug: doxorubicin hydrochloride
Drug: prednisone
Drug: vincristine sulfate
Radiation: yttrium Y 90 ibritumomab tiuxetan

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as doxorubicin, vincristine, and cyclophosphamide, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Steroid therapy, such as prednisone, may be effective in treating cancer and blocking the body's immune response. Monoclonal antibodies, such as rituximab and yttrium Y 90 ibritumomab tiuxetan, can block cancer growth in different ways. Some block the ability of cancer cells to grow and spread. Others find cancer cells and help kill them or carry cancer-killing substances to them. Giving chemotherapy together with prednisone and monoclonal antibody therapy may kill more cancer cells.

PURPOSE: This phase II trial is studying how well giving doxorubicin together with vincristine, cyclophosphamide, prednisone, and rituximab followed by rituximab and yttrium Y 90 ibritumomab tiuxetan works in treating patients with newly diagnosed large B-cell lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine event-free survival of patients with large B-cell lymphoma treated with CHOP-R followed by consolidation therapy.

Secondary

* Determine overall survival.
* Evaluate relapse-free survival for patients achieving complete or partial response.
* Determine the rate of disease progression.
* Determine response rate at the end of study therapy.
* Assess the toxicities of this regimen.

OUTLINE: This is a multicenter study.

* Induction therapy: Patients receive the CHOP-R regimen comprising doxorubicin hydrochloride IV, vincristine IV, cyclophosphamide IV, and rituximab IV on day 1 and prednisone IV on days 1-5. Treatment repeats every 2 weeks for 2 courses.

Patients who achieve complete or partial response, as assessed by PET/CT scan, receive a third course of induction therapy.

* Consolidation therapy: Patients receive rituximab IV on days -8 to 0 and yttrium Y 90 ibritumomab tiuxetan IV on day 0.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed large B-cell lymphoma

  * Stage I, II, III, or IV disease
  * Bone marrow or lymph node involvement by small cell lymphoma allowed
  * No serious, progressive pathology (at investigator's discretion)
* CD20-positive disease
* Measurable disease
* No prior indolent lymphoma, treated or not
* No meningeal or CNS lymphoma

PATIENT CHARACTERISTICS:

* International prognostic index < 2 (adjusted for age)
* Life expectancy > 3 months
* ALT and AST ≤ 2.5 times upper limit of normal
* Bilirubin ≤ 30 mmol/L
* Creatinine ≤ 150 μmol/L
* HIV, hepatitis B virus, and hepatitis C virus negative (unless after vaccine)
* No contraindication to chemotherapy or immunotherapy
* No cancer in the past 5 years except basal cell skin cancer or carcinoma in situ of the cervix
* No contraindication to a venous catheter

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* At least 30 days since prior and no other concurrent investigational treatment
* No prior therapy
* No concurrent participation in another clinical study

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 30 (Actual)
Dates: Start 2007-05; Primary Completion 2010-03 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Event-free survival | 1 year

SECONDARY OUTCOMES:
Overall survival | up to one year
Relapse-free survival in responding patients | up to one year
Rate of disease progression | up to 2 years
Response rate | up to six months
Toxicities | up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Frederec Peyrade, MD, Study Chair — Centre Antoine Lacassagne
Locations (1):
- Centre Antoine Lacassagne, Nice, France